CLINICAL TRIAL: NCT04370899
Title: Early Detection of Familial Hypercholesterolemia in Children in Tarragona Province
Brief Title: Early Detection of Familial Hypercholesterolemia in Children
Acronym: DECOPIN
Status: Recruiting | Type: Observational
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Principal Investigator, Nuria Plana, Principal Investigator, Institut Investigacio Sanitaria Pere Virgili
Other Study IDs: 176/2018
Record Dates: First submitted 2020-02-28; First posted 2020-05-01 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Familial Hypercholesterolemia; Familial Hypercholesterolemia - Heterozygous; Familial Hypercholesterolemia - Homozygous
Keywords: Familial Hypercholesterolemia; Childhood; cardiovascular risk; lifestyle assessment; genetic disorder; LDL cholesterol
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Homozygous Familial Hypercholesterolemia; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Familial hypercholesterolaemia children: FH diagnostic criteria were as follows: a positive genetic test or, if no genetic test results were available, LDL-C >160 mg/dL and one parent with a DLCN score >8.
  Interventions: Other: lifestyle assessment
- Unaffected children: The children evaluated for suspected FH who did not meet the FH criteria were included in the non-FH control group
  Interventions: Other: lifestyle assessment

INTERVENTIONS:
Other: lifestyle assessment — A semi-quantitative assessment of the consumption of different food groups will be carried out using a frequency questionnaire validated by the Spanish population27. This questionnaire consists of 137 food items and will be obtained by the dietitian of our Unit (see annex).
  The child population and/or their parents will be instructed on how to fill the data in the food diary for a period of 3 days, in order to be able to analyse the nutritional composition of the intake and the effect on the lipid profile. The first food register, will be obtained at the collection visit before starting any type of treatment. Another food diary will be included after one year.
  Physical activity will be collected from the Minnesota Test and we will ask about the consumption of tobacco.

SUMMARY:
Heterozigous FH is an underdiagnosed disease in the paediatric population. Its early detection, would allow us to initiate lifestyle therapeutical changes and early pharmacological therapy if necessary. This is a key fact to reduce atherosclerosis progression and cardiovascular risk in adulthood. Moreover, it will allow, detecting the first and second degree affected relatives.

DETAILED DESCRIPTION:
The most prevalent cause of hypercholesterolemia in childhood is Heterozygous Familial Hypercholesterolemia (HeFH).

It is a monogenic disorder that is transmitted of autosomal dominant way and affects 50% of offspring. It is characterized by the increase of low-density lipoproteins (LDL-C), which can be detected from birth. It is mostly caused by mutations in the gene that encodes the LDL receptor (LDLr) located in the short arm of chromosome 19. Nowadays, more than 1500 different mutations have been described worldwide. Less common are the ApoB3500 Family Defect, caused by the mutation of the Apolipoprotein B gene (APOB) that is located on chromosome 2, and the mutation of the gene encoding PCSK9 (proprotein convertase subtilisin-kexin type 9) located on the chromosome 1p32.2. These three entities are clinically expressed in the same way and only the genetic study will allow us to differentiate them.

HeFH has a prevalence of 1 for every 250 individuals in the European population, therefore it is the most frequent genetic disease, which is a major public health problem as it is associated with high cardiovascular risk (CVR). In spite of the current knowledge and the diagnostic techniques, it continues being an unknown disease and therefore is underdiagnosed and under-treated. In countries with active screening projects of HeFH detection, only 20% are diagnosed. In Catalonia, in order to get free access to lipid lowering therapy, a register was started in 2004. In November 2012, a total of 2,981 patients were registered in Catalonia, representing 19.53% of expected HeFH patients in Catalonia. Only 108 children were included, in the age group 0 to 14 years, In clinical practice, DLCN criteria (clinical criteria of Dutch Lipids Units) is used as a diagnostic tool, but these clinical criteria cannot be applied to the children. The criteria are based on family history, personal history, physical examination and LDL-C levels. A definite clinical diagnosis of HeFH is considered when the score obtained is equal to or greater than 8 points, it´s probable when the score obtained is between 6-7 points and possible when it is between 3-5 points (table 1). In these clinical criteria, the presence of tendinous xanthomas and the corneal arch are very important. These two stigmas are not present in HeFH children, and the investigators will only find xanthomas in Homozygous Familial Hypercholesterolemia (HoFH). This form of the disease is very serious and the prevalence is low, 1 per 300,000-400,000 habitants.

It suspect HeFH when the investigators observe LDL levels >135 mg/dL in children with a family history of premature cardiovascular disease (men < 55 y/o and women < 65 y/o) in first-degree relatives, or a parent with LDL levels> 240 mg/dL (according to data published in adult HeFH population in the Spanish population).

At present, there are clear evidences that high LDL-C levels in children induce the formation and development of atheromatous lesion. This lesion can be initiated during the first years of life by cholesterol deposit, causing an increase in the carotid intimate-medium thickness (cIMT), progressing silently until adulthood.

It has been observed in children over 5 years of age that high cholesterol levels cause alterations in endothelial function of the arterial wall, measured by flow-mediated dilation (FMD). Wigman and colleagues observed that cIMT of HeFH children between 8 - 18 years H was higher than the control children population, estimating cIMT growth in around 0.0047 mm/year; in front of 0.0003 mm/year in the control group. Dalmau and colleagues evaluated the cIMT of 88 HeFH children between 2 and 19 years and described a faster cIMT increase with age particularly after 12 years old, regardless of gender and other analytical parameters related to CVR.

Statin intervention studies, have described that reductions between 30 and 40% in LDL-C levels lead to an improvement in endothelial function measured by FMD and cIMT. It has also observed that arterial stiffness was increased in children with CVR compared to children without CVR.

There is evidence suggesting that HeFH children have a pro-inflammatory and pro-oxidant state that could accelerate the atherosclerosis process and increase CVR. Recent studies from our group have shown that E-selectin, sVCAM or oxLDL/LDL are associated with lower post-ischemia reactivity in small arteries in patients with high CVR.

Statin intervention studies in HeFH children have proven that these drugs are safe and effective. LDL-C reduction is associated to a reduction in cIMT. An early lipid lowering therapy decrease the lifelong CVR.

The first clinical guidelines addressing familial hypercholesterolemia (FH) in children were published in 1992 by National Cholesterol Education Program (NCEP). Since then, many Scientific Societies have given recommendations about detection, diagnosis and treatment. All guides reinforce the importance of an early detection. The most conflicting point between the different panels of experts is the type of screening. The National Heart Lung and Blood Institute (NHLBI) recommends universal screening between 9 and 11 years, in the context of the comprehensive management of CVR factors in childhood, and selective screening between 2 and 8 years. Other guidelines recommend selective screening based on family history and the presence of CVR factors.

A recent study has shown that screening based on lipid profile may be insufficient to detect HeFH population. A genetic study of 215 members of 24 families with RLDL mutations showed that 7% of the members wear the mutation despite a normal lipid profile.

The Netherlands is one of the countries with a more active health policies to detect the HeFH population. For many years, they have established a National Program based in cascade screening of all first-degree relatives of diagnosed FH patients. They propose a general screening of the children population between 1 and 9 years. This type of screening has a greater sensitivity and specificity. Universal screening together with selective screening would be the most efficient method to detect FH patients, but this goal can only be achieved by activating specific healthcare strategies in the usual clinical practice.

One group of investigators assessed the degree of control and follow-up of 207 HeFH children (0-18 y/o) from January 2007 to May 2008. Only 62% had received a lifestyle change advice,16% took functional foods every day with stanols or sterols and only 26% were taking statin therapy. Their conclusions were that a screening program is necessary but this programme should be accompanied by a proper follow-up with a multidisciplinary health group (nurses, pediatricians, dietitians and specialists involved in the management of severe hypercholesterolemia).

Previously, different studies had observed that 50% of men and 20% of woman with FH don't received adequate treatment increasing the risk of coronary episodes before 50 years old. Nowadays, it has been shown that the intensive treatment of FH patients reduce cardiovascular mortality, reaching the same proportion as the general population.

According the official data from the "Generalitat of Catalonia" the province of Tarragona has a population of 71,186 children between the ages of 0 and 14. The aim of this project is detecting FH children early to improve their CVR in adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Children between 2 and 18 years of age.
* LDL-C level above 135 mg/dL
* Previously, the pediatrician will have discarded secondary causes (hypercholesterolaemia such as hypothyroidism, nephrotic syndrome, diabetes, renal insufficiency).

After confirmation that one of the parents has a genetic mutation (Lipoxip/Liponext) or clinical diagnosis (DLCN ≥ 8), the child will be studied. The progenitor with hypercholesterolemia will be considered as an index case, in this way we will demonstrate the vertical transmission of the genetic disease.

Exclusion Criteria:

* The child population under 2 and over the age of 18 and children.
* Children with high cholesterol but by secondary causes.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between 2 and 18 years of age who have a LDL-C level above 135 mg/dL.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-03-14 (Actual); Primary Completion 2030-03-14 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Number the children detected of FH | From date of randomization until the date of first documented progression, assessed up to 10 years.
  The main result of the study is to increase the number of children affected by FH, as well as to detect their families.

SECONDARY OUTCOMES:
LDL-cholesterol level (mg/dl) at entry and at follow-up | every year, up to 10 years
  LDL-cholesterol measurement at enrolment and after follow-up.
Healthy habits of population | every year, up to 10 years
  Food frequency questionnarie will be carried out by a registered dietician-nutritionist every year to see if children improve their diet

CONTACTS AND LOCATIONS:
Overall Officials: Luis Masana, MD, PhD, Study Director — Institut Investigacio Sanitaria Pere Virgili
Locations (2):
- Spain (2):
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital Universitari Sant Joan, Reus, Tarragona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Plana N, Rodriguez-Borjabad C, Ibarretxe D, Masana L. Familial hypercholesterolemia in childhood and adolescents: A hidden reality. Clin Investig Arterioscler. 2017 May-Jun;29(3):129-140. doi: 10.1016/j.arteri.2016.11.002. Epub 2017 Apr 5. English, Spanish. PMID 28390853
- [Result] Rodriguez-Borjabad C, Malo AI, Ibarretxe D, Girona J, Heras M, Ferre R, Feliu A, Salvado M, Varela A, Amigo N, Masana L, Plana N; DECOPIN Group; DECOPIN GROUP Investigators who have participated in patient recruitment. Efficacy of therapeutic lifestyle changes on lipid profiles assessed by NMR in children with familial and non-familial hypercholesterolemia. Clin Investig Arterioscler. 2020 Mar-Apr;32(2):49-58. doi: 10.1016/j.arteri.2019.10.001. Epub 2020 Jan 29. English, Spanish. PMID 32005605
- [Result] Ibarretxe D, Rodriguez-Borjabad C, Feliu A, Bilbao JA, Masana L, Plana N. Detecting familial hypercholesterolemia earlier in life by actively searching for affected children:The DECOPIN project. Atherosclerosis. 2018 Nov;278:210-216. doi: 10.1016/j.atherosclerosis.2018.09.039. Epub 2018 Oct 1. PMID 30312929
- [Result] Plana N, Rodriguez-Borjabad C, Ibarretxe D, Ferre R, Feliu A, Caselles A, Masana L; en representacion del proyecto DECOPIN. Lipid and lipoprotein parameters for detection of familial hypercholesterolemia in childhood. The DECOPIN Project. Clin Investig Arterioscler. 2018 Jul-Aug;30(4):170-178. doi: 10.1016/j.arteri.2017.12.003. Epub 2018 Mar 27. English, Spanish. PMID 29602595
- [Result] Rodriguez-Borjabad C, Ibarretxe D, Girona J, Ferre R, Feliu A, Amigo N, Guijarro E, Masana L, Plana N; DECOPIN Group. Lipoprotein profile assessed by 2D-1H-NMR and subclinical atherosclerosis in children with familial hypercholesterolaemia. Atherosclerosis. 2018 Mar;270:117-122. doi: 10.1016/j.atherosclerosis.2018.01.040. Epub 2018 Jan 31. PMID 29407879

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT04370899/Prot_SAP_000.pdf